CLINICAL TRIAL: NCT04241484
Title: Piezowave Myofascial Acoustic Compression Therapy on Lateral and Medial Tendinopathies
Brief Title: Piezowave for Treatment on Lateral and Medial Elbow Tendinopathies
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00237364
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Elbow Tendinopathy; Golfer's Elbow; Medial Epicondylitis; Lateral Epicondylitis; Tennis Elbow
MeSH Terms: conditions — Elbow Tendinopathy; Tennis Elbow

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Piezowave (Experimental): * Initiation of Piezowave MyACT treatment to include parameters from the user manual
  * Set for frequency of five pulses per second
  * Delivery of 500 to 1000 pulses over multiple injured area sites, not to exceed 4000 pulses per session
  * Intensity ranging from 0.1 to 18 millijoule per square millimeter. This intensity if energy flux as the rate of transfer of the energy through the surface of the tissue is applied.
  * Focal transducer
  * Head size will be variable based on depth of tissue treated. The user manual will be consulted for depth of penetration recommendations
  Interventions: Device: Piezowave 2

INTERVENTIONS:
Device: Piezowave 2 — Piezowave Myofascial Acoustic Compression Therapy (MyACT), which provides mechanical stimuli delivery to improve circulation and provide relief of pain. The focused sound waves produced by the Piezowave MyACT device are classified by a pressure surge, which is followed by a drop in pressure and a brief negative pressure phase low energy/low pressure application. It is this transformation of mechanical stimuli into biochemical signals, or mechanotransduction, which yields the treatment of myofascial and musculoskeletal pain

SUMMARY:
Within the outpatient rehabilitation clinic, therapists provide therapeutic interventions to treat patients with various tendinopathies, including lateral and medial epicondylosis. Current conservative treatment includes immobilization for forced rest of the inflamed tendons and muscles, as well as mobilizations to focus stimulation of synovial fluid, provide movement to nourish cartilage, promote periarticular extensibility, and provide sensory and proprioceptive input. Musculoskeletal disorders can accompany both local and referred pain patterns that need to be assessed and treated. When an acute trauma or repetitive micro-trauma occurs, that may result in decreased range of motion and increased pain causing the onset of weakness and function of the affected extremity. An alternative approach is through the provision of Piezowave Myofascial Acoustic Compression Therapy (MyACT), which provides mechanical stimuli delivery to improve circulation and provide relief of pain. The focused sound waves produced by the Piezowave MyACT device are classified by a pressure surge, which is followed by a drop in pressure and a brief negative pressure phase low energy/low pressure application. It is this transformation of mechanical stimuli into biochemical signals, or mechanotransduction, which yields the treatment of myofascial and musculoskeletal pain. There is currently limited research to support the benefit in regards to increased function and decreased pain when the Piezowave MyACT is used for the treatment of lateral and medial epicondylosis. Of the limited research available, treatment with non-invasive shock wave therapy, complications are low and effect is achieved in most cases within three to five sessions.

If Piezowave Myofascial Acoustic Compression Therapy (MyACT)) is applied as treatment for symptoms of lateral and medical elbow tendinopathies, then the patient will experience increased function demonstrated by Quick DASH (Disability of the Arm, Shoulder and Hand) score and decreased pain demonstrated by subjective reporting on the numeric pain rating scale.

ELIGIBILITY:
Inclusion Criteria:

* Tendinopathy symptoms referred for occupational therapy by physician.
* Positive provocation tests

Exclusion Criteria:

* Contraindications for shock wave

  * Infections
  * Tumor tissue
  * Blood clotting disorder
  * Blood thinning medication use
  * Pregnancy
  * Lung tissue in focal area
  * Head
  * Air-containing organs
  * Elbow fracture
* History of corticosteroid injections less than eight weeks/two months, prior to initiation of occupation therapy treatment for lateral or medial epicondylosis. The goal would be to have elimination of any residual benefit from the injection.

Ages: 22 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Function as demonstrated by Quick score | The Quick score will be completed by the participant at the initial evaluation or session and repeated at visit 10 or at day 30 day post-intervention, which ever comes first.
  The Quick (Disability of the Arm, Shoulder and Hand) score will assess participant report of function based on daily activities by creating an upper extremity functional score. There are 11 questions that ask the participant to rate their difficulty or limitations and pain in order to complete specific tasks. Each questions will ask the participant to select one of the five measures from no difficulty, not limited at all or none to unable, extreme and I can't sleep, with the latter of the measures indicating decreased upper extremity function. A maximum total score of 55 and minimum of 11.

SECONDARY OUTCOMES:
Change in Pain level as demonstrate by the numeric pain rating scale | The participant will be asked to report their pain will be completed by the participant at the initial evaluation or session and repeated at visit 10 or at day 30 day post-intervention, which ever comes first.
  The participant will document their pain level as assessed by the numeric pain rating scale from 0 to 10. 0 represents no pain and 10 represents the greatest level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Christa Schestag, MSOT, Principal Investigator — Outpatient Rehabilitation Services

IPD SHARING:
Plan to Share IPD: No